CLINICAL TRIAL: NCT01330888
Title: Exploring Deployment Stress and Reintegration in Army National Guard Chaplains
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: D7800-P
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Combat Stress Disorder
Keywords: war; religion; caregiver; combat stress disorder
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: ARNG Chaplains

SUMMARY:
The purpose of this 2-year pilot study is to explore the impact of deployment on the psychosocial and health characteristics and reintegration of Military Chaplains, specifically those of the Army National Guard (ARNG). This pilot will serve as the foundation for subsequent investigations of chaplains from multiple branches of the military. In addition to spiritual and religious support, Military Chaplains play a key role in the behavioral health of deployed service-members, routinely participating in suicide prevention training, conducting critical event debriefing, and identifying service-members at risk for combat and operational stress reactions1. A high risk group for exposure to trauma2, Military Chaplains have suffered brain injuries, gunshot wounds and blast injuries in OEF/OIF Theater3. In addition, many report combat related stress issues such as compassion fatigue, PTSD, and reintegration issues3. While the traumatic experiences of OEF/OIF deployed troops have been well documented, the effects on military chaplains caring for these service-members have received little attention in the research to date. We are collaborating with the National Guard Chaplain Corps Leadership on this program of research. The aims of this 2-year pilot cross-sectional study focus on describing and exploring deployment and its impact on psychosocial, health characteristics and reintegration of ARNG chaplains using a mixed method approach (web-based survey, in-depth interviews, social network analysis).

ELIGIBILITY:
Inclusion Criteria:

* current, active members of ARNG during timeframe of OIF/OEF/OND
* Chaplains
* able to be contacted by email for survey explanation and participation
* consent to participate in interview or network questionnaire

Exclusion Criteria:

* not current, active members of ARNG during timeframe of OIF/OEF/OND
* not Chaplains
* not able to be contacted by email for survey explanation and participation
* do not consent to participate in interview or network questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ARNG Chaplains who have ever/never been deployed to OEF/OIF combat theaters
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
observational | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen Besterman-Dahan, PhD MA BS, Principal Investigator — James A. Haley Veterans' Hospital
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, Florida, United States

REFERENCES:
- [Result] Besterman-Dahan K, Barnett S, Hickling E, Elnitsky C, Lind J, Skvoretz J, Antinori N. Bearing the burden: deployment stress among army national guard chaplains. J Health Care Chaplain. 2012;18(3-4):151-68. doi: 10.1080/08854726.2012.723538. PMID 23094615
- [Result] Besterman-Dahan K, Gibbons SW, Barnett SD, Hickling EJ. The role of military chaplains in mental health care of the deployed service member. Mil Med. 2012 Sep;177(9):1028-33. doi: 10.7205/milmed-d-12-00071. PMID 23025131